CLINICAL TRIAL: NCT03117790
Title: Impact of Dexmedetomidine Supplemented Analgesia on Sleep Quality in Elderly Patients After Major Surgery: A Randomized, Double-blind, and Placebo-controlled Pilot Study
Brief Title: Impact of Dexmedetomidine on Sleep Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman,Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEXsleep
Record Dates: First submitted 2017-04-02; First posted 2017-04-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Elderly; Surgery; Analgesia; Dexmedetomidine; Complication,Postoperative; Sleep Quality
Keywords: elderly; surgery; analgesia; dexmedetomidine; sleep quality
MeSH Terms: conditions — Agnosia; Postoperative Complications; Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Morphine (0.5 mg/ml, in a total volume of 160 ml) is used for patient-controlled analgesia. Dexmedetomidine (200 ug) is added to the formula of patient-controlled analgesia. Patient-controlled analgesia is provided during the first 3 days after surgery.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Morphine (0.5 mg/ml, in a total volume of 160 ml) is used for patient-controlled analgesia. Placebo (normal saline) is added to the formula of patient-controlled analgesia. Patient-controlled analgesia is provided during the first 3 days after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Morphine (0.5 mg/ml, in a total volume of 160 ml) is used for patient-controlled analgesia. Dexmedetomidine (200 ug) is added to the formula of patient-controlled analgesia. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time from 6 to 8 minutes.
  Other Names: Dexmedetomidine supplemented morphine analgesia
  Arms: Dexmedetomidine group
Drug: Placebo — Morphine (0.5 mg/ml, in a total volume of 160 ml) is used for patient-controlled analgesia. Placebo (normal saline) is added to the formula of patient-controlled analgesia. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time from 6 to 8 minutes.
  Other Names: Morphine analgesia
  Arms: Placebo group

SUMMARY:
Sleep disturbances frequently occur in elderly patients after major surgery; and their occurrence are associated with worse outcomes including increased incidence of delirium. Previous studies showed that, for elderly patients admitted to the ICU after non-cardiac surgery, low-dose dexmedetomidine infusion improved to some degree the quality of sleep and reduced the incidence of delirium. The investigators hypothesize that, for elderly patients after major non-cardiac surgery, dexmedetomidine supplemented analgesia can also improve the sleep quality. The purpose of this randomized controlled pilot study is to investigate the impact of dexmedetomidine supplemented analgesia on the sleep quality in elderly patients after major non-cardiac surgery.

DETAILED DESCRIPTION:
Sleep disturbances usually develop in elderly patients after major surgery, which are manifested as prolonged sleep latencies, shortened sleep duration, frequent wake-up, disordered circadian rhythm, abnormally increased stages 1 and 2 non-rapid eye movement (N1 and N2) sleep, and decreased or absent slow wave sleep (SWS) and rapid eye movement (REM) sleep. Occurrence of sleep disturbances is harmful for the recovery of both physiological and mental functions after surgery, and may even lead to the development of postoperative complications. For example, study showed that postoperative sleep disturbances were associated with increase risks of delirium, cardiovascular events and infections, prolonged durations of stay in ICU and hospital, increased medical expenses and high mortality rate. However, methods that may effectively improve the quality of postoperative sleep are still lacking.

Multiple factors are responsible for the development of sleep disturbances after surgery. These include (1) environmental factors, such as noises, lights, medical and nursing activities, etc.; (2) comorbid diseases, such as cardiovascular disease, inflammatory reaction, infections, etc.; (3) stress response and pain stimulation provoked by surgery, especially major surgery; (4) mechanical ventilation. Studies found significantly disordered circadian rhythms, fragmented sleep and absent REM sleep in mechanically ventilated patients; and (5) multiple medications, such as benzodiazepines, opioids, non-steroidal anti-inflammatory drugs, and glucocorticoids,.

Dexmedetomidine is a high selective alpha 2 adrenoceptor agonist which produces hypnosis and sedation by activating the alpha 2 adrenoceptor in the locus coeruleus of the brain; it is well known that the locus coeruleus is the key part to adjust sleep and awakening. The study of Nelson et al. showed that dexmedetomidine induces the expression of c-Fos in the locus coeruleus nucleus and ventral lateral nucleus in rats' brain, which is similar to the expression of c-Fos during non-rapid eye movement sleep. They presumed that dexmedetomidine activates the endogenous sleep-promoting pathway to produce sedative effects, which is totally different from benzodiazepines and opiates on the mechanism.

A recent study of the investigators showed that, in elderly patients who were admitted to the ICU after surgery and did not require mechanical ventilation, low-dose dexmedetomidine infusion (at a rate of 0.1 ug/kg/h, for 15 hours) prolonged the total sleep time, increased the percentage of N2 sleep (and reduced the percentage of N1 sleep), increased the efficiency of sleep and improved the subjective sleep quality. Another study of the investigators showed that low-dose dexmedetomidine infusion in elderly patients who were admitted to the ICU after non-cardiac surgery improved the subjective sleep quality and reduced the daily prevalences of delirium during the first 3 days after surgery. We hypothesize that dexmedetomidine supplemented analgesia can improve the structure and circadian rhythm of sleep, and reduce the incidence of delirium in elderly patients after major non-cardiac surgery.

Simple randomization was performed. Random numbers were generated in a 1:1 ratio with a block size of 4 using the SAS 9.2 software (SAS Institute, USA). Study drugs (either 200 μg/2 ml dexmedetomidine hydrochloride or 2 ml 0.9% saline) were provided as clear aqueous solution in the same type of 3 ml volume ampules (manufactured by Jiangsu Hengrui Medicine Co, Ltd, China) and encoded according to the randomization results before the study by a pharmacist who did not participate in the rest of the study. The results of randomization were sealed in sequentially numbered envelopes until the end of the study.

Dexmedetomidine was not permitted in either group. Anesthesia was induced with midazolam (0.02-0.03 mg/kg), propofol, and sufentanil. Muscle relaxation was achieved using rocuronium, under some special circumstances, using succinylcholine or awake intubation is feasible. Anesthesia was maintained with a propofol infusion and sufentanil or remifentanil, as well as cis-atracurium, rocuronium, with or without the volatile anesthetic sevoflurane or the inhaled gas nitrous oxide. The Bispectral Index were adjusted between 40 and 60. The Bispectral Index is an electroencephalographic measure of hypnotic depth, which ranging from 0 to 100, with values between 40 and 60 considered optimum.

Sequential randomization numbers were assigned to vials by a pharmacist who was otherwise not involved in the trial. All investigators, clinicians, and patients were therefore completely blinded to treatment allocation. But in case of emergency (such as unexpected, rapid deterioration in a participant's clinical status), clinicians could adjust or stop drug administration if deemed clinically necessary. Unmasking was not allowed unless clearly needed for clinical purposes.

Postoperative analgesia was provided with a patient-controlled intravenous analgesia of the trial drug (either dexmedetomidine 200 μg or 0.9% saline) and 80 mg morphine, diluted with 0.9% saline to 160 ml. The patient-controlled pump was programmed to deliver 2-mL boluses with a lockout interval of 8 minutes and a background infusion at 1 mL/h. We adopt this dosing regimen because it has been safely used in our clinical practice and our previous studies. Patient-controlled analgesia was continued for at least 24 h, but not longer than 72 h after surgery. Other analgesics including non-steroidal anti-inflammatory drugs, acetaminophen, and opioids were administered when considered necessary. Open-label dexmedetomidine was not allowed except for treatment of delirium.

Patients were transferred to the post-anesthesia care unit and remained for at least 30 min, monitoring non-invasive blood pressure, electrocardiogram, and pulse oxygen saturation. Then they were sent to a surgical ward. Non-invasive blood pressure and pulse oxygen saturation were monitored intermittently until next morning. Non-invasive blood pressure and heart rate were then monitored once or twice daily until hospital discharge. Those who were unstable were monitored more frequently and transferred to an intensive care unit for clinical purposes. For postoperative patient who accidently came to the intensive care unit, polysomnography monitoring would not be performed.

Polysomnography was performed with a SOMNO watch plus (SOMNO medics GmbH, Germany) from 9:00 PM on the day of surgery until 6:00 AM on the first day after surgery. Two qualified investigators (Z.-F.Z. and X.-Q.M.) were responsible for attaching the electrodes to the patients. The polysomnogram included six-channel electroencephalogram (F3, F4, C3, C4, O1, O2), two-channel electrooculogram (EOG) and one-channel chin electromyogram (EMG). These data were processed according to the American cademy of Sleep Medicine manual (AASM)automatically and stored safely in a research computer disc. A qualified sleep physician who was blinded to the study protocol and did not participate in data collection and patient care scored the sleep architecture epoch by epoch by using the American cademy of Sleep Medicine manual. Total sleep architecture was divided into wakefulness, NREM sleep (stage 1, stage 2, and stage 3), and REM sleep. Total sleep time was defined as the sum of time spent in any sleep stage during the monitoring period. Sleep efficiency was calculated as the ratio between the total sleep time and the total recording time and expressed as percentage. The percentages of each sleep stage were calculated as the durations of each sleep stage divided by the total sleep time. Sleep fragmentation index was calculated as the average number of arousals and awakenings per hour.

Research staffs were blind to randomization, and were not permitted to communicate with either patients or their doctors about any group assignment or treatment. These who responsible for postoperative assessments was not allowed to participate in anesthesia and perioperative care of patients.

Baseline data included demographic characteristics, surgical diagnosis, pre-operative comorbidities, surgical history, smoking and alcohol consumption, and pre-operative medications and laboratory test results and the Charlson Comorbidity Index. Cognitive function was evaluated with the Mini-Mental State Examination (MMSE), score ranges from 0 to 30, with higher score indicating better function. Sleep quality was evaluated with the Pittsburgh Sleep Quality Index, score ranges from 0 to 21, with higher score indicating worse sleep quality. Subjective sleep quality (Refer to the Richards Campbell sleep scale, a 11-point scale where 0 indicates the best possible sleep and 10 indicates the worst possible sleep) and Pain intensity (A 11-point scale where 0 indicates no pain and 10 indicates the worst pain) were also evaluated. Routine intraoperative monitoring included electrocardiogram, non-invasive blood pressure, pulse oxygen saturation, end-tidal carbon dioxide, volatile anesthetic concentration, and urine output. Intra-arterial pressure and central venous pressure were monitored only if necessary. Postoperative data included, study drug and morphine consumption during patient-controlled analgesia, supplemental analgesics and hypnotics within 5 days, and other medications.

All enrolled patients were assessed twice daily, between 8:00-10:00 AM and 6:00-8:00 PM, until the 5th postoperative day or hospital discharge or death, whichever occurred first. Subjective sleep quality was recorded with Numeric Rating Scale (NRS, an 11-point scale where 0=the best sleep and 10=the worst sleep). Sedation level was assessed using the RASS (Richmond Agitation-Sedation Scale), with scores ranging from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm. If RASS score reached -4 or -5, which meant the patients were extremely sedated or unconsciousness. Delirium was not assessed. Delirium was assessed with CAM-ICU (Confusion Assessment Method for the Intensive Care Unit). Delirium was classified into three motoric subtypes: (1) hyperactive (RASS score was consistently positive, +1 to +4); (2) hypoactive (RASS score was consistently neutral or negative, -3 to 0); and, (3) mixed.

Other prespecified outcomes included postoperative pain intensity both at rest and with movement, which was assessed twice daily at the time of delirium with Numeric Rating Scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) during the first 5 postoperative days; adverse events from the beginning of patient-controlled analgesia until 72 hours after surgery; postoperative complications within 30 days; 30-day mortality; 30 days after surgery. By using Chinese version Telephone Interview for Cognitive Status-modified (TICS-m; scores ranging from 0 to 48, with higher scores indicating better cognitive function), the cognitive function was assessed. Quality-of-life was assessed with the World Health Organization Quality of Life-brief version, (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. The score of each domain ranges from 0 to 100, with higher score indicating better function).

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 65 years
2. Scheduled to undergo elective non-cardiac major surgery (with expected duration >= 2 hours) under general anesthesia
3. Transferred to general ward with a patient-controlled intravenous analgesia pump after surgery.

Exclusion Criteria:

1. Refuse to participate
2. Preoperative history of schizophrenia, epilepsy, parkinsonism or myasthenia gravis
3. Patients with preoperative sleep disorders (accepted sedatives or hypnotics within 1 month before surgery) or the STOP-BANG Questionnaire score is 3 or higher
4. Inability to communicate in the preoperative period because of coma, profound dementia or language barrier
5. Brain injury or neurosurgery
6. Preoperative left ventricular ejection fraction < 30%, sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker
7. Severe hepatic dysfunction (Child-Pugh class C); Severe renal dysfunction (requirement of renal replacement therapy before surgery); ASA classification IV or unlikely to survive for more than 24 hours after surgery
8. Patients recruited in other studies
9. Other conditions that are considered unsuitable for study participation

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
The percentage of stage N2 sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring

SECONDARY OUTCOMES:
The duration of stage N1 sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The percentage of stage N1 sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The duration of stage N2 sleep | During the night after surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The duration of stage N3 sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The percentage of stage N3 sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The duration of REM sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
The percentage of REM sleep | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Determined by polysomnographic monitoring
Total sleep time | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Total time spent in any sleep stage during the monitoring period. Determined by polysomnographic monitoring.
Sleep efficiency | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  The ratio between the total sleep time and the total recording time and expressed as percentage. Determined by polysomnographic monitoring.
Sleep fragmentation index | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  The average number of arousals and awakenings per hour of sleep. Determined by polysomnographic monitoring

OTHER OUTCOMES:
Pain intensity | Up to the fifth day after surgery
  Estimated with numeric rating scale, where 0 = no pain and 10 the most severe pain
Subjective sleep quality | Up to the fifth day after surgery
  Estimated with numeric rating scale, where 0 = the best sleep and 10 the worst sleep.
Sedation level | Up to the fifth day after surgery
  Assessed using the Richmond Agitation-Sedation Scale (RASS), with scores ranging from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm.
Cumulative consumption of morphine | Up to the fifth day after surgery
  Cumulative morphine consumption after surgery
Incidence of delirium | During the first 5 days after surgery
  Incidence of delirium within 5 days after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of postoperative complications | Up 30 days after surgery
  Incidence of non-delirium complications within 30 days after surgery
30-day mortality | On the 30th day after surgery
  All cause mortality on the 30th day after surgery
Quality of life | On the 30th day after surgery
  Quality of life is assessed with the World Health Organization Quality of Life-brief version (WHOQOL-BREF; a 24-item questionnaire that provides assessments of the quality of life in 4 domains. The score of each domain ranges from 0 to 100, with higher score indicating better function).
Cognitive function | On the 30th day after surgery
  Cognitive function is assessed with the Telephone Interview for Cognitive Status-modified (TICS-m; score ranges from 0 to 50, with higher score indicating better function).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drouot X, Roche-Campo F, Thille AW, Cabello B, Galia F, Margarit L, d'Ortho MP, Brochard L. A new classification for sleep analysis in critically ill patients. Sleep Med. 2012 Jan;13(1):7-14. doi: 10.1016/j.sleep.2011.07.012. Epub 2011 Dec 6. PMID 22153778
- [Background] Gabor JY, Cooper AB, Hanly PJ. Sleep disruption in the intensive care unit. Curr Opin Crit Care. 2001 Feb;7(1):21-7. doi: 10.1097/00075198-200102000-00004. PMID 11373507
- [Background] Figueroa-Ramos MI, Arroyo-Novoa CM, Lee KA, Padilla G, Puntillo KA. Sleep and delirium in ICU patients: a review of mechanisms and manifestations. Intensive Care Med. 2009 May;35(5):781-95. doi: 10.1007/s00134-009-1397-4. Epub 2009 Jan 23. PMID 19165463
- [Background] Stanchina ML, Abu-Hijleh M, Chaudhry BK, Carlisle CC, Millman RP. The influence of white noise on sleep in subjects exposed to ICU noise. Sleep Med. 2005 Sep;6(5):423-8. doi: 10.1016/j.sleep.2004.12.004. Epub 2005 Mar 31. PMID 16139772
- [Background] Salas RE, Gamaldo CE. Adverse effects of sleep deprivation in the ICU. Crit Care Clin. 2008 Jul;24(3):461-76, v-vi. doi: 10.1016/j.ccc.2008.02.006. PMID 18538195
- [Background] Kamdar BB, Needham DM, Collop NA. Sleep deprivation in critical illness: its role in physical and psychological recovery. J Intensive Care Med. 2012 Mar-Apr;27(2):97-111. doi: 10.1177/0885066610394322. Epub 2011 Jan 10. PMID 21220271
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Weinhouse GL, Schwab RJ, Watson PL, Patil N, Vaccaro B, Pandharipande P, Ely EW. Bench-to-bedside review: delirium in ICU patients - importance of sleep deprivation. Crit Care. 2009;13(6):234. doi: 10.1186/cc8131. Epub 2009 Dec 7. PMID 20053301
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Schiza SE, Simantirakis E, Bouloukaki I, Mermigkis C, Arfanakis D, Chrysostomakis S, Chlouverakis G, Kallergis EM, Vardas P, Siafakas NM. Sleep patterns in patients with acute coronary syndromes. Sleep Med. 2010 Feb;11(2):149-53. doi: 10.1016/j.sleep.2009.07.016. Epub 2010 Jan 18. PMID 20083431
- [Background] Friese RS. Sleep and recovery from critical illness and injury: a review of theory, current practice, and future directions. Crit Care Med. 2008 Mar;36(3):697-705. doi: 10.1097/CCM.0B013E3181643F29. PMID 18176314
- [Background] Friese RS, Diaz-Arrastia R, McBride D, Frankel H, Gentilello LM. Quantity and quality of sleep in the surgical intensive care unit: are our patients sleeping? J Trauma. 2007 Dec;63(6):1210-4. doi: 10.1097/TA.0b013e31815b83d7. PMID 18212640
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Fanfulla F, Ceriana P, D'Artavilla Lupo N, Trentin R, Frigerio F, Nava S. Sleep disturbances in patients admitted to a step-down unit after ICU discharge: the role of mechanical ventilation. Sleep. 2011 Mar 1;34(3):355-62. doi: 10.1093/sleep/34.3.355. PMID 21358853
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Weinhouse GL, Watson PL. Sedation and sleep disturbances in the ICU. Crit Care Clin. 2009 Jul;25(3):539-49, ix. doi: 10.1016/j.ccc.2009.04.003. PMID 19576529
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Derived] Zhang ZF, Su X, Zhao Y, Zhong CL, Mo XQ, Zhang R, Wang K, Zhu SN, Shen YE, Zhang C, Wang DX. Effect of mini-dose dexmedetomidine supplemented intravenous analgesia on sleep structure in older patients after major noncardiac surgery: A randomized trial. Sleep Med. 2023 Feb;102:9-18. doi: 10.1016/j.sleep.2022.12.006. Epub 2022 Dec 20. PMID 36587547